CLINICAL TRIAL: NCT03598257
Title: A Phase II Randomized Trial of Olaparib (NSC-747856) Administered Concurrently With Radiotherapy Versus Radiotherapy Alone for Inflammatory Breast Cancer
Brief Title: Radiation Therapy With or Without Olaparib in Treating Patients With Inflammatory Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01519; NCI-2018-01519 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S1706 (Other: SWOG); S1706 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2018-07-24; First posted 2018-07-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Breast Inflammatory Carcinoma
Keywords: Inflammatory breast cancer; Olaparib; Radiation therapy
MeSH Terms: conditions — Inflammatory Breast Neoplasms | interventions — Specimen Handling; olaparib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (olaparib, radiation therapy) (Experimental): Patients receive olaparib PO BID the day before standard RT commences (Day 0) and throughout the RT course until the last day of RT administration. Olaparib is also continued on weekends (routine days without RT) throughout the RT course. Patients undergo standard radiation therapy 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Olaparib; Radiation: Radiation Therapy; Other: Survey Administration
- Group II (radiation therapy) (Active Comparator): Patients undergo standard radiation therapy 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Radiation: Radiation Therapy; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281
  Arms: Group I (olaparib, radiation therapy)
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Other: Survey Administration — Ancillary study

SUMMARY:
This phase II trial studies how well radiation therapy with or without olaparib works in treating patients with inflammatory breast cancer. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Olaparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy. It is not yet known whether radiation therapy with or without olaparib may work better in treating patients with inflammatory breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the invasive disease-free survival (IDFS) of patients with inflammatory breast cancer receiving concurrent administration of olaparib with standard doses of radiotherapy to the chest wall and regional lymph nodes compared to standard doses of radiotherapy alone to the chest wall and regional lymph nodes.

SECONDARY OBJECTIVE:

I. To compare the effect of concurrent administration of olaparib with radiotherapy versus radiotherapy alone on improvement in locoregional control (measured by locoregional recurrence-free interval), distant relapse-free survival, and overall survival in inflammatory breast cancer patients.

ADDITIONAL OBJECTIVE:

I. To collect tissue and whole blood for processing and banking in anticipation of future correlative studies in this patient population.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive olaparib orally (PO) twice daily (BID) the day before standard radiation therapy (RT) commences (Day 0) and throughout the RT course until the last day of RT administration. Olaparib is also continued on weekends (routine days without RT) throughout the RT course. Patients undergo radiation therapy 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients undergo standard radiation therapy 5 days per week for 6 weeks in the absence of disease progression or unacceptable toxicity.

Patients undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up within 5 weeks, then every 3 months until 3 years after registration, and then every 6 months for up to 8 years after registration.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have inflammatory breast cancer without distant metastases. All biomarker subtype groups (estrogen receptor [ER], progesterone receptor [PR], HER2) are eligible. Inflammatory disease will be defined per American Joint Committee on Cancer (AJCC) 8th edition with documentation by history/exam and pathology at the time of diagnosis.
* All patients must have completed neoadjuvant chemotherapy prior to mastectomy. The chemotherapy regimen is at the discretion of the treating physician but it is recommended that it include at least 4 cycles of anthracycline and/or taxane-based therapy (plus targeted therapy for patients with HER2+ disease). Response to chemotherapy is not a criterion for eligibility (both complete responders and those with residual disease are eligible). Please note that although pathologic complete response (pCR) is not required or excluded, pCR status must be determined post-surgery prior to randomization.
* All patients must have undergone modified radical mastectomy (with negative margins on ink) with pathologic nodal evaluation (from level I and II axillary lymph node dissection [ALND]) at least 3 weeks and no more than 12 weeks prior to randomization, unless they receive additional chemotherapy after mastectomy. Patients must not have gross residual tumor or positive microscopic margins after mastectomy.
* Additional adjuvant chemotherapy after surgery is allowed at the discretion of the treating physician, either completed prior to randomization or planned for after completion of protocol treatment. If adjuvant chemotherapy is administered after mastectomy, the patient must be randomized at least 3 weeks but no more than 12 weeks after the last dose of adjuvant chemotherapy.
* Patients must not have a history of radiation therapy to the ipsilateral chest wall and/or regional nodes. Prior radiation therapy to other body sites is allowed.
* Patients must not be planning to receive any other investigational agents during radiation therapy. Prior therapy, including prior treatment with olaparib or other PARP inhibitor, is allowed.
* Patients must not have a known hypersensitivity to olaparib or any of the excipients of the product.
* Patients must not have unresolved or unstable grade 2 or greater toxicity (with the exception of alopecia) from prior administration of another investigational drug and/or prior anti-cancer treatment.
* Patients must not be planning to receive strong or moderate CYP3A inhibitors or inducers while on olaparib treatment. Patients receiving strong or moderate CYP3A inhibitors must agree to discontinue use at least 2 weeks prior to receiving olaparib. Patients receiving strong or moderate CYP3A inducers must agree to discontinue use at least 5 weeks prior to receiving olaparib.
* Patients must not be planning to receive live virus or live bacterial vaccines while receiving olaparib and during the 30 day follow up period
* Patients must not be planning to receive any additional anti-cancer therapy (chemotherapy, endocrine therapy, immunotherapy, biological therapy or other novel agent) while receiving radiotherapy with or without study medication. If a patient is receiving concurrent anti-HER2 targeted therapies, they must not take these medications during the period of radiotherapy (with or without study drug) while enrolled on the study.
* Patients must be >= 18 years of age
* Patients must have Zubrod performance status 0-2.
* Absolute neutrophil count (ANC) >= 1000/mm^3 (within 28 days prior to registration)
* Platelet count >= 100,000/mm^3 (within 28 days prior to registration)
* Hemoglobin >= 9.0 g/dL (after transfusion if required and within 28 days prior to registration)
* Patients must have adequate renal function as evidenced by calculated creatinine clearance >= 51 mL/min by Cockcroft-Gault equation, within 28 days prior to registration.
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 28 days prior to registration)

  * Patients with documented Gilbert's disease may have bilirubin up to 2.5 mg/dL
* Serum glutamic-oxaloacetic transaminase (SGOT) =< 2.5 x ULN (within 28 days prior to registration)
* Serum glutamate pyruvate transaminase (SGPT) =< 2.5 x ULN (within 28 days prior to registration)
* Alkaline phosphatase =< 2.5 x ULN (within 28 days prior to registration)
* Patients must not have a history of other prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for five years
* Female patients must be postmenopausal or have a negative urine or serum pregnancy test within 14 days prior to registration. Female patients of childbearing potential (and male patients with female partners who are of childbearing potential or pregnant) who are sexually active, must agree to the use of two highly effective forms of contraception during protocol treatment and for 6 months following the last dose of olaparib. Note: The efficacy of hormonal contraceptives may be reduced if co-administered with olaparib. Male patients must agree not to donate sperm during protocol treatment and for 6 months after the last dose of olaparib.
* Patients who are breastfeeding must agree to discontinue breastfeeding before receiving olaparib due to potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib.
* Patients must not have active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Patients must be able to swallow and retain oral medications and have no known gastrointestinal disorders likely to interfere with absorption of the study medication.
* Patients must not have a history of a resting electrocardiography (ECG) indicating uncontrolled, potentially reversible cardiac conditions (such as unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, Fridericia's formula corrected QT interval [QTcF] prolongation > 500 ms, electrolyte disturbances) or congenital long QCYP3T syndrome.
* Patients must not have myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Patient must not have had major surgery within 2 weeks of starting study treatments and patients must have recovered from any effects of any major surgery.
* Patients must not have a history of uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan.
* Patients must not have had previous allogenic bone marrow transplant or double umbilical cord blood transplantation (dUCBT).
* Patients must not have had whole blood transfusions in the last 120 days prior to randomization.
* Patients must be offered the opportunity to participate in specimen submission for banking.

  * Note: Germline and somatic BRCA status (genetic testing) are planned for future correlative evaluation, in order to examine treatment and circulating tumor deoxyribonucleic acid (ctDNA) response as stratified by BRCA 1/2 mutational status. Since this is future planned correlative research, any mutational status results would not be returned to the patient or the treating physician. There is no Clinical Laboratory Improvement Act (CLIA)-certified clinical genetic testing being performed for patients as part of the S1706 study. A forthcoming revision or separate corelative sciences proposal would be submitted to and approved by National Cancer Institute (NCI) prior to conduct of any planned future translational medicine objectives.
* Patients who can complete the patient-reported outcomes (PRO) Quality of Life (QOL) and PRO-CTCAE questionnaires in English must be offered the opportunity to participate in the optional PRO substudy. Patients who are not able to complete questionnaires in English need not be offered the opportunity to participate.
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.
* As a part of the OPEN registration process, the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (IDFS) | Up to 8 years
  Time from date of registration to date of first invasive recurrence (local, regional or distant), second invasive primary cancer (breast or not), or death due to any cause. Patients last known to be alive who have not experienced recurrence or second primary cancer are censored at their last contact date. Analysis will be on an intent-to-treat basis and will estimate the survival endpoints using the product-limit method of Kaplan-Meier and will compare the time-to-event distributions using log-rank test statistics. Hazard ratios will be calculated from Cox regression analyses. Effect modification by the stratification variables will be tested as interactions with treatment and separate hazard ratios with 95% confidence intervals by major subgroups will be displayed in a forest plot to examine for consistency of the treatment effect over these subgroups.

SECONDARY OUTCOMES:
Locoregional Recurrence-Free Interval (Local Disease-Free Interval [LDFI]) | Up to 8 years
  Time from date of registration to date of invasive local or regional recurrence. Patients last known to be alive without recurrence are censored at their last contact date. Patients with distant recurrence, second primary cancer or death are censored at the time of that event. A competing risk framework will be conducted separating out the event types of locoregional recurrence from distant recurrence and death. Hazard ratios will be calculated from Cox regression analyses. Effect modification by the stratification variables will be tested as interactions with treatment and separate hazard ratios with 95% confidence intervals by major subgroups will be displayed in a forest plot to examine for consistency of the treatment effect over these subgroups.
Distant Relapse-Free Survival (Distant Recurrence-Free Survival) | Up to 8 years
  Time from date of registration to date of invasive distant disease recurrence, second invasive primary cancer (breast or not) or death due to any cause. Patients last known to be alive who have not experienced disease recurrence, or second primary cancer are censored at their last contact date.
Overall Survival | Up to 8 years
  Time from date of registration to date of death due to any cause. Patients last known to be alive are censored at their last contact date.

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Jagsi, Principal Investigator — SWOG Cancer Research Network
Locations (220):
- United States (214):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - NEA Baptist Memorial Hospital and Fowler Family Cancer Center - Jonesboro, Jonesboro, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Shaw Cancer Center, Edwards, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Beebe South Coastal Health Campus, Millville, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - TidalHealth Nanticoke / Allen Cancer Center, Seaford, Delaware
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - IU Health West Hospital, Avon, Indiana
  - IU Health North Hospital, Carmel, Indiana
  - IU Health Central Indiana Cancer Centers-Fishers, Fishers, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - IU Health Methodist Hospital, Indianapolis, Indiana
  - McFarland Clinic - Ames, Ames, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Ascension Via Christi Hospitals Wichita, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - University Medical Center New Orleans, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Corewell Health Dearborn Hospital, Dearborn, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Henry Ford Health Providence Novi Hospital, Novi, Michigan
  - Michigan Healthcare Professionals Pontiac, Pontiac, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Henry Ford Health Providence Southfield Hospital, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Gulfport Memorial Hospital, Gulfport, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Capital Health Medical Center-Hopewell, Pennington, New Jersey
  - Valley Health System Ridgewood Campus, Ridgewood, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Lovelace Radiation Oncology, Albuquerque, New Mexico
  - Memorial Medical Center-Las Cruces, Las Cruces, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Pluta Cancer Center, Rochester, New York
  - University of Rochester, Rochester, New York
  - Mission Hospital, Asheville, North Carolina
  - Hope Women's Cancer Centers-Asheville, Asheville, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - UH Seidman Cancer Center at Firelands Regional Medical Center, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - University Hospitals Sharon Health Center, Wadsworth, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cancer Centers of Southwest Oklahoma Research, Lawton, Oklahoma
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - MD Anderson in The Woodlands, Conroe, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - MD Anderson West Houston, Houston, Texas
  - Doctor's Hospital of Laredo, Laredo, Texas
  - MD Anderson League City, League City, Texas
  - MD Anderson in Sugar Land, Sugar Land, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - United Hospital Center, Bridgeport, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - ThedaCare Regional Cancer Center, Appleton, Wisconsin
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Canada (4):
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - CHU de Quebec-L'Hotel-Dieu de Quebec (HDQ), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Puerto Rico (2):
  - San Juan Community Oncology Group, San Juan
  - Centro Comprensivo de Cancer de UPR, San Juan

REFERENCES:
- [Derived] Michmerhuizen AR, Pesch AM, Moubadder L, Chandler BC, Wilder-Romans K, Cameron M, Olsen E, Thomas DG, Zhang A, Hirsh N, Ritter CL, Liu M, Nyati S, Pierce LJ, Jagsi R, Speers C. PARP1 Inhibition Radiosensitizes Models of Inflammatory Breast Cancer to Ionizing Radiation. Mol Cancer Ther. 2019 Nov;18(11):2063-2073. doi: 10.1158/1535-7163.MCT-19-0520. Epub 2019 Aug 14. PMID 31413177